CLINICAL TRIAL: NCT06872346
Title: Personalized Risk-based Follow-up of Cervical Cancer Screening in Practice (PREDICT), Randomized Control Trial
Brief Title: Personalized Risk-based Follow-up of Cervical Cancer Screening in Practice, RCT
Acronym: PREDICT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer S Haas, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 24-646
Record Dates: First submitted 2025-02-28; First posted 2025-03-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical Cancer; Screening; Clinical Decision Support
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Control Arm (Standard Care) patients will receive the usual care provided by their PCP, practice, and/or specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Standard Care (No Intervention): Patients will receive the usual care provided by their PCP, practice, and/or specialist.
- Arm 2: Visit Based Reminder (Active Comparator): Visit based reminders for physicians and patients that will be seen in Epic and Patient Gateway
  Interventions: Other: Visit-based IT reminders to patients and practitioners
- Arm 3: Population Health Outreach (Active Comparator): Visit based reminders for physicians and patients that will be seen in Epic and Patient Gateway. Patients will received outreach from a population health coordinator. Patients will be sent educational materials, a reminder letter, and if needed, additional help scheduling their follow up appointment.
  Interventions: Other: Visit-based IT reminders to patients and practitioners; Other: Population outreach

INTERVENTIONS:
Other: Visit-based IT reminders to patients and practitioners — To identify patients due for CCSM, simplify test ordering/referral, and track follow-up, PREDICT will include: 1) automated updating of a patient's problem list with the current cervical screening finding, 2) automated updating of cervical cancer health maintenance topics to the appropriate time interval and follow-up test/ procedure through the use of modifiers, 3) "SmartSets" to standardize ordering of procedures/ specialty referrals.
  Arms: Arm 2: Visit Based Reminder; Arm 3: Population Health Outreach
Other: Population outreach — Patients will be sent a reminder letter 90 days prior to the due date via the patient portal or mailed if no portal account (Outreach 1). If needed, four weeks later a phone call from the outreach coordinator reminds patients of the follow-up date if scheduled or helps establish follow-up (Outreach 2). The coordinator could also place an order for a referral and send a reminder to the practitioner to sign it if appropriate. The coordinator will review and document any "alternative care plans" discussed by the PCP and patient.
  Arms: Arm 3: Population Health Outreach

SUMMARY:
The goal of this PREDICT is to assess a personalize approach to screening and management of cervical cancer testing. The investigators will evaluate patients who are due for a follow up cervical cancer screening in the primary care clinics in the Massachusetts General Brigham system. Patients will be randomized by clinic into three different arms (Arm 1: standard care, Arm 2: visit based reminders, Arm 3: visit based reminders and population health outreach)

DETAILED DESCRIPTION:
Cancer screening and management guidelines are moving from a "one size fits all" approach to one that is tailored to an individual. Cervical Cancer Screening Management (CCSM) is the first example of a guideline that incorporates longitudinal screening history to personalize risk assessment. While a personalized approach offers the promise of enhancing the balance of benefits vs. harms of screening and management, this ideal can only be realized through strong systems to support care delivery. Without IT tools that integrate personalized algorithms with care delivery, more errors of judgement may occur if practitioners and patients are confused about appropriate next steps. The investigators hypothesize that delivering risk based CCSM to all eligible individuals will require: 1) using a generalizable Clinical Decision Support (CDS) tool that is validated and open source to implement the American Society for Colposcopy and Cervical Pathology (ASCCP) recommendations; 2) leveraging a system level health IT platform to present risk-based, personalized recommendations; and 3) offering a stepped care approach that individually engages patients and primary care physicians (PCP); and 4) enhances team-functioning, with increasing intensity over time (Figure 1). Accordingly, the investigators propose to develop, implement, and rigorously test PREDICT (Personalized Risk-based Follow-up of Cervical Cancer Screening in Practice) within 4 primary care practice networks.

PREDICT components include supporting individual patient and practitioner engagement, and enhancing team coordination through an efficient "stepped care" approach. This will be compared to standard care by the patient's care team using a 3-arm, randomized design that will allow us to examine the marginal and cumulative effectiveness of the intervention components.

The study will be conducted in four primary care networks that are part of a large healthcare system (Mass General Brigham [MGB]): two affiliated with academic medical centers (Brigham and Women's Hospital [BWH] and Massachusetts General Hospital [MGH]), and two affiliated with community hospitals (Newton Wellesley Hospital [NWH] and North Shore Medical Center [NSMC])

PREDICT will include multilevel components. These will be tested using the 3-arm design that allows assessment of the sequential addition of these components. This design will also evaluate changing the responsibility for "opportunistic" follow-up, typically by the practitioner or patient at the time of a visit, to a systematic, multilevel approach, examining the cumulative and marginal effects of each subsequent level of intervention. In addition to the multilevel components, the individual- and team-level engagement algorithm will take a "stepped care" approach with increasing level of intensity of engagement

Step 1 will start 90 days before the date an individual is due for follow-up ("due date"), at the time of enrollment, based on the patient's personalized risk score. For example, Step 1 for a patient with a 5-year CIN 3+ risk of 0.6% in a practice randomized to an intervention arm would automatically have a 1-year surveillance follow-up reminder set in the EHR. In these intervention practices, practitioners could access this information when in the patient's EHR or when the patient views the reminder in their patient portal. For practices randomized to Arm 3, Step 2 would begin with a patient being sent a reminder letter 90 day prior the due date via the patient portal or mailed if no portal account (Outreach 1). If needed, four weeks later a phone call from the outreach coordinator reminds patients of the follow-up date if scheduled or helps establish follow-up (Outreach 2). The coordinator could also place an order for a referral and send a reminder to the practitioner to sign it if appropriate. The coordinator will review and document any "alternative care plans" discussed by the PCP and patient. A SQL study database will include functionality for coordinators to know when a patient should be contacted, how many contacts have been made, and the outcome of those efforts. Intervention components in Arm 3 will differ for individuals recommended for 3-year surveillance and for individuals 65 years and older who have prior abnormalities that would warrant additional surveillance or diagnostic management. In Arm 3, individuals recommended for 3-year surveillance will only receive Outreach 1 reminder letters (the study will have insufficient resources to make phone calls). Since individuals 65 years and older who have prior abnormalities that would warrant additional surveillance or diagnostic management are more likely to have other comorbid conditions that may affect recommended follow-up, study coordinators will message practitioners prior to performing patient outreach.

ELIGIBILITY:
Inclusion Criteria, Individuals who:

* have a cervix and are 21-70 years old
* receive care at a participating primary care practice (i.e. PCP team visit within past 3 years)
* have had a Pap and/ or HPV test within the past 3.5 years
* has a CCSM result that suggest a 5-year risk of developing CIN3+ that warrants surveillance at 1 or 3 years, diagnostic colposcopy, or treatment (i.e., above average risk).

Inclusion of those up to age 70 is intended to identify individuals whose prior history does not meet screening exit criteria, and warrants surveillance or diagnostic care even though women with adequate prior screening can stop at age 65

Exclusion Criteria Individuals who:

* were diagnosed with cervical cancer/ CIN3+ prior to the most recent screening Pap or HPV test
* have had their cervix removed
* are not English or Spanish-speaking.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness outcome | 120 days
  The primary effectiveness outcome, measured at the patient level, is receipt of follow-up within 120 days of the due date, extracted from EHR/ associated claims documentation, for individuals with a 5-year risk of developing CIN3+ of 0.6% or more. This time interval was selected to allow patients sufficient time to move through the stepped care intervention with enough time to schedule recommended follow-up given practitioner availability

SECONDARY OUTCOMES:
Secondary effectiveness outcome | 240 days
  The secondary effectiveness outcome, number of days to completion over a 240 day follow-up period, to examine whether follow-up occurs as quickly as possible with censoring at the end of study period for patients who never receive follow-up.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT06872346/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT06872346/SAP_001.pdf